CLINICAL TRIAL: NCT03666793
Title: Comprehensive Management of Drug Prescriptions Throughout the Elderly Person's Hospital Care, From Hospital to Home: Impact on Readmission at 30 Days After Delivery
Brief Title: Comprehensive Management of Drug Prescriptions Throughout the Elderly Person's Hospital Care
Acronym: OPTISORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC-P0069
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Elderly; Medication Reconciliation; Patient Readmission
Keywords: Elderly; Medication Reconciliation; Patient Readmission
MeSH Terms: interventions — Quality Indicators, Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard healthcare procedures
- experimental: Reconciliation group (Experimental): medical reconciliation at admission, multidisciplinary medication review, medical reconciliation at discharge of the hospital
  Interventions: Other: global care

INTERVENTIONS:
Other: global care — Medication Reconciliation at admission, Multidisciplinary medication review, Medication Reconciliation at discharge
  Arms: experimental: Reconciliation group

SUMMARY:
This study evaluates the impact of optimizing drug prescriptions on re-admissions of elderly patients within 30 days after hospital discharge. It compares a group of patients receiving comprehensive care (medication reconciliation at hospital entry, multidisciplinary medication review, and medication reconciliation at discharge), versus another group that does not benefit from the program.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in the department of short geriatric stay

Exclusion Criteria:

* Patients already included in the study, and readmitted in the same service.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2019-01-17 (Actual)

PRIMARY OUTCOMES:
Rate of readmission at 30 days | 30 days
  Evaluate the impact of optimizing drug prescriptions on re-admissions of elderly patients within 30 days of return to home.Only direct re-admissions to emergency and geriatric short-stay services in participating centres will be counted.

SECONDARY OUTCOMES:
Time between discharge and first readmission | 30 days
  Evaluate the impact of medication management on the time required for the first re-admission to hospital, if it takes place before 30 days.
Rate of changes in the prescription after hospital discharge by the general practitioner | 30 days
  Estimate the impact of this process on the preservation of the prescription after hospital discharge by general practitioner within the 30 days following the return home actual number of discrepancies, what may have caused the change and which are the concerned drugs
Identification of Seniors at Risk (ISAR) score | 30 days
  This score is based on 6 yes/no questions. T e total scale range is from 0 to 6. Each item is scored 1 if there is a problem or 0 if there is not, being the maximum score =6.

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Visade, MD, Principal Investigator — GHICL
Locations (1):
- GHICL, Lomme, France